CLINICAL TRIAL: NCT06560333
Title: Evaluate the Efficacy and Safety of the Combined Use of a Sodium-glucose Cotransporter 2 (iSGLT2) Inhibitor and a Dipeptidyl Peptidase-4 (iDPP -4) Inhibitor in the Treatment of Type 2 Diabetes Mellitus in Patients Treated With Metformin
Brief Title: iSGLT2 Inhibitor and a iDPP -4 Inhibitor in Treatment of Type 2 Diabetes Mellitus in Patients Treated With Metformin (TRIAD)
Acronym: TRIAD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic change in development priorities
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF186
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N0892 (Experimental): in the test group will be required to take 3 tablet of the test drug N0892. 3 tablets a day for 84 days +/- 4 days.
  Interventions: Drug: N0892
- Forxiga® + Glifage XR® + Placebo of Januvia® (Active Comparator): in the control group will be required to take 1 tablet of Forxiga® 10mg, 1 tablet of Glifage XR® 1000mg and 1 tablet of Placebo of Januvia® 100mg. 3 tablets a day for 84 days +/- 4 days.
  Interventions: Drug: Forxiga® + Glifage XR® + Placebo
- Januvia® + Glifage XR® + Placebo of Forxiga® (Active Comparator): in the control group will be required to take 1 tablet of Januvia® 100mg, 1 tablet of Glifage XR® 1000mg and 1 tablet of Placebo of Forxiga® 100mg. 3 tablets a day for 84 days +/- 4 days.
  Interventions: Drug: Januvia® + Glifage XR® + Placebo

INTERVENTIONS:
Drug: N0892 — 1 tablet of Forxiga® 10mg, 1 tablet of Januvia® 100mg and 1 tablet of Glifage XR® 1000mg
  Arms: N0892
Drug: Januvia® + Glifage XR® + Placebo — 1 tablet of Januvia® 100mg, 1 tablet of Glifage XR® 1000mg and 1 tablet of Placebo of Forxiga ®10mg
  Arms: Januvia® + Glifage XR® + Placebo of Forxiga®
Drug: Forxiga® + Glifage XR® + Placebo — 1 tablet of Forxiga ®10mg, 1 tablet of Glifage XR® 1000mg and 1 tablet of Placebo of Januvia ® 100mg
  Arms: Forxiga® + Glifage XR® + Placebo of Januvia®

SUMMARY:
The present study aims to evaluate the efficacy and safety of different combinations of oral antidiabetics in patients with inadequate glycemic control on metformin monotherapy.

DETAILED DESCRIPTION:
This is a phase III, multicenter, randomized, double-blind, double-dummy clinical trial to evaluate the efficacy and safety of the he fixed-dose combination in patients diagnosed with type 2 DM (Diabetes mellitus), with or without cardiovascular or renal complications, and who did not reach the therapeutic goals of glycemic control with previous guidance on diet and physical exercise, on monotherapy with metformin at the maximum tolerated dose, and who, at the discretion of the Investigator, may benefit from the addition of trial drugs.

The trial will have a total duration of a maximum of 144 days (approximately 20 weeks), with a screening/run-in period of up to 4 weeks and 16 weeks (112 ± 4 days) of treatment. The trial will include a screening visit (V-1), a baseline randomisation visit (V0), three follow-up visits (V1, V2, V3) and a final visit (V4).

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree with all the purposes of the trial, signing and dating the ICF in two copies;
* Age equal to or over 18 years old and less than or equal to 80 years old
* Diagnosis of type 2 DM with uncontrolled glycemia with a history of HbA1c ≥7.5% and ≤10.5% (up to 12 previous months) with previous guidance on diet and physical exercise and monotherapy with metformin at the maximum tolerated dose (≥1,000 mg/day, stable and without signs of intolerance in the last 12 weeks) and who, at the Investigator's discretion, may benefit from the addition of the trial drugs

Exclusion Criteria:

* Any clinical observation finding (clinical/physical assessment) or laboratory condition that is interpreted by the investigating physician as a risk to the research Subject's participation in the clinical trial or the presence of uncontrolled chronic disease(s);
* History of alcohol or illicit drug use disorder in the two years prior to the Visit;
* Subjects who are pregnant, breastfeeding or planning to become pregnant, or female subjects of childbearing potential who are not using a reliable method of contraception;
* Known history of allergy or hypersensitivity to any of the trial treatments, or to the excipients in the formulas, or in case of rare hereditary diseases which may be incompatible with the excipients in the product formulas (such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption);
* Subjects with type 1 diabetes mellitus;
* History of fasting blood glucose ≥ 270 mg/dL.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-11-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the glycemic control at week 16 | 16 weeks
  Evaluate the superiority of the combined use of N0892 in glycemic control (reduction in HbA1c: Glycated haemoglobin) at week 16 in subjects receiving metformin, compared to Forxiga® and Januvia® alone

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil